CLINICAL TRIAL: NCT00143247
Title: An Open-Label, Phase 2, Long-Term Safety Study of Inhaled Insulin: An Up to Four-Year Extension of Therapy in Subjects With Type 1 or Type 2 Diabetes Mellitus Participating in Extension Protocols 217-102, 103, or 104
Brief Title: Long-Term Safety Study of Inhaled Insulin: An Up to Four-Year Extension of Therapy in Subjects With Type 1 or Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2171036
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2009-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exubera® (inhaled insulin) (Experimental): Open label, no comparator
  Interventions: Drug: Exubera® (inhaled insulin)

INTERVENTIONS:
Drug: Exubera® (inhaled insulin) — Treatment of type 1 and type 2 diabetes with short-acting insulin
  Other Names: Exubera®

SUMMARY:
This is a long-term safety study for Phase 2 subjects who choose to remain on Exubera® (inhaled insulin).

DETAILED DESCRIPTION:
The study was terminated on Oct. 18, 2007. This study is not a post approval commitment study. Pfizer decided to cancel new trials because of the decision to withdraw Exubera® (inhaled insulin) due to lack of market performance and not for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 1 or Type 2 Diabetes Mellitus who participated in previous Phase 2 extension protocols

Exclusion Criteria:

* Smoking
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2003-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171036&StudyName=An%20Optional%20Roll-Over%20Extension%20of%20Previous%20Phase%202%20Available%20to%20Patients%20Who%20Participated%20in%20Previous%20Phase%202%20Studies.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with type 1 or 2 diabetes in 1 of parent Phase 2 protocols (217-102,103,or 104)& received EXUBERA® (EXU)were enrolled. 173 subjects were screened,assigned to treatment,and treated for at least 1 day.For each subject,data from controlled and extension studies were combined to represent each subject's entire EXU exposure experience.
Pre-assignment Details: The objective of the study was to observe,in subjects with long-term exposure to EXUBERA®,pulmonary function over time.For each subject,data from the controlled study (217-102,103,and 104) were combined with data from the respective extension studies as well as the A2171036 extension study to represent each subject's entire EXU exposure experience.
Groups:
- Inhaled Insulin: Open label EXUBERA® (EXU; inhaled insulin), no comparator. At all times in the trial, each subject had an individualized recommended insulin dose for each of the dosing times. Initial recommended doses for EXU were based on the subject's weight, any previous responses to insulin, and other factors noted in the protocol.
Period: Overall Study
Arm/Group | Inhaled Insulin
Started | 173 (173=total subjects of current + 3 previous protocols)
Completed | 17
Not Completed | 156
Not completed — Death | 8
Not completed — Adverse Event | 19
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 55
Not completed — Study terminated by sponsor | 31
Not completed — Protocol Violation | 15
Not completed — Lost to Follow-up | 12
Not completed — following inaccurate lab adverse event | 1
Not completed — Other | 12

BASELINE CHARACTERISTICS:
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 173
Age Continuous [Mean (Standard Deviation); unit: years] | 46.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 103

OUTCOME MEASURES:

1. Secondary Outcome: Change in Glycosylated Hemoglobin by Duration of Exubera Treatment
Description: Change from Baseline: mean of (value of observed glycosylated hemoglobin (HbA1C) (percent) at treatment duration minus baseline value). Duration of treatment is based on the elapsed duration of treatment in the controlled and uncontrolled studies. Baseline was based on pre-inhaled insulin measurements.
Time Frame: Baseline to 126 months
Population: 173 subjects received at least one treatment. The safety analysis set (subjects who received at least one dose of EXU treatment) were included in analysis. n = subjects who had outcome measure data available at particular time points. There was no imputation for missing data.
Measure: Mean (Standard Deviation); unit: percent HbA1C
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 157
percent HbA1C
  3 months (n=155) | -0.99 (1.37)
  6 months (n=146) | -0.90 (1.58)
  12 months (n=136) | -0.60 (1.72)
  18 months (n=121) | -0.66 (1.61)
  24 months (n=115) | -0.65 (1.67)
  30 months (n=107) | -0.67 (1.72)
  36 months (n=99) | -0.60 (1.73)
  42 months (n=93) | -0.61 (1.72)
  48 months (n=88) | -0.48 (1.64)
  54 months (n=83) | -0.50 (1.61)
  60 months (n=75) | -0.48 (1.56)
  66 months (n=70) | -0.56 (1.82)
  72 months (n=67) | -0.61 (1.87)
  78 months (n=62) | -0.80 (1.47)
  84 months (n=57) | -0.71 (1.26)
  90 months (n=56) | -0.75 (1.51)
  96 months (n=54) | -0.58 (1.46)
  102 months (n=50) | -0.77 (1.52)
  108 months (n=42) | -0.68 (1.51)
  114 months (n=37) | -0.78 (1.60)
  120 months (n=31) | -0.39 (1.46)
  126 months (n=23) | -0.08 (1.22)

2. Secondary Outcome: Hypoglycemic Event Rates by Interval of Exubera Treatment
Description: Number of hypoglycemic events per subject-month. Subject-month determined by time on treatment. Interval of treatment based on elapsed duration of treatment in the controlled & uncontrolled studies.Overall represents entire duration of treatment. Hypoglycemia: Characteristic symptoms of hypoglycemia with no blood glucose check. Clinical picture must include prompt resolution with food intake, subcutaneous glucagon or intravenous glucose.OR,Characteristic symptoms of hypoglycemia with blood glucose check showing glucose <=59 mg/dl.OR,Any glucose measurement <=49 mg/dl,with or without symptoms.
Time Frame: 0 to 132 months
Population: as for outcome 1
Measure: Number; unit: events / subject-month
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 159
events / subject-month
  0 to 4 weeks (n=159) | 2.38
  >4 to 8 weeks (n=158) | 2.10
  >8 to 12 weeks (n=157) | 1.92
  >12 weeks to 6 months (n=155) | 1.88
  >6 to12 months (n=149) | 1.91
  >12 to18 months (n=134) | 1.63
  >18 to 24 months (n=122) | 1.96
  >24 to 30 months (n=112) | 1.99
  >30 to 36 months (n=107) | 1.78
  >36 to 42 months (n=98) | 1.54
  >42 to 48 months (n=91) | 1.47
  >48 to 54 months (n=85) | 1.36
  >54 to 60 months (n=80) | 1.38
  >60 to 66 months (n=74) | 1.32
  >66 to 72 months (n=70) | 1.42
  >72 to 78 months (n=64) | 1.47
  >78 to 84 months (n=59) | 1.74
  >84 to 90 months (n=58) | 1.63
  >90 to 96 months (n=56) | 1.67
  >96 to 102 months (n=52) | 1.52
  >102 to 108 months (n=48) | 1.16
  >108 to 114 months (n=40) | 1.51
  >114 to 120 months (n=37) | 1.41
  >120 to 126 months (n=25) | 1.13
  >126 to 132 months (n=18) | 0.92
  Overall (n=159) | 1.65

3. Secondary Outcome: Severe Hypoglycemic Event Rates by Interval of Exubera Treatment
Description: Number of severe hypoglycemic events per 100 subject-months.Subject-month determined by time on treatment.Interval of treatment based on elapsed duration of treatment in controlled & uncontrolled studies.Overall represents entire duration of treatment.A severe hypoglycemic event must have met all 3of following:1.subject unable to treat self.2.subject exhibited 1 or more of neurological symptoms defined in protocol.3.blood glucose must be <=49 mg/dl if measured.If not measured,clinical manifestations must have been reversed by oral carbohydrates,subcutaneous glucagon,or intravenous glucose.
Time Frame: 0-132 months
Population: as for outcome 1
Measure: Number; unit: severe events / 100 subject-months
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 159
severe events / 100 subject-months
  0-4 weeks (n=159) | 1.37
  >4-8 weeks (n=158) | 2.76
  >8-12 weeks (n=157) | 0.70
  >12 weeks-6months (n=155) | 2.64
  >6-12 months (n=149) | 1.07
  >12-18 months (n=134) | 0.93
  >18-24 months (n=122) | 0.85
  >24-30 months (n=112) | 1.07
  >30-36 months (n=107) | 0.97
  >36-42 months (n=98) | 0.18
  >42-48 months (n=91) | 0.19
  >48-54 months (n=85) | 0.60
  >54-60 months (n=80) | 0.87
  >60-66 months (n=74) | 0.47
  >66-72 months (n=70) | 0.75
  >72-78 months (n=64) | 0.27
  >78-84 months (n=59) | 1.14
  >84-90 months (n=58) | 1.47
  >90-96 months (n=56) | 0.31
  >96-102 months (n=52) | 1.32
  >102-108 months (n=48) | 0.39
  >108-114 months (n=40) | 0.44
  >114-120 months (n=37) | 0.54
  >120-126 months (n=25) | 0
  >126-132 months (n=18) | 0
  Overall (n=159) | 0.88

4. Secondary Outcome: Insulin Antibodies (Percent Binding) by Time on Exubera Treatment - Subjects With Type 1 Diabetes
Description: Observed values by duration of treatment.
Time Frame: 36 months to 126 months
Population: as for outcome 1
Measure: Median (Full Range); unit: percent binding
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 61
percent binding
  36 months (n=31) | 26.00 (23.95) [1.50 to 88.00]
  42 months (n=4) | 27.00 (15.44) [4.00 to 37.00]
  48 months (n=28) | 19.00 [1.50 to 64.00]
  54 months (n=27) | 16.00 [1.50 to 63.00]
  60 months (n=26) | 14.00 [1.50 to 83.00]
  66 months (n=23) | 16.00 [1.50 to 66.00]
  72 months (n=22) | 13.00 [1.50 to 81.00]
  78 months (n=24) | 14.00 [3.00 to 84.00]
  84 months (n=23) | 16.00 [1.50 to 67.00]
  90 months (n=21) | 13.00 [1.50 to 77.00]
  96 months (n=23) | 18.00 [1.50 to 77.00]
  102 months (n=21) | 14.00 [1.50 to 76.00]
  108 months (n=17) | 18.00 [1.50 to 83.00]
  114 months (n=15) | 11.00 [1.50 to 65.00]
  120 months (n=14) | 8.50 [1.50 to 75.00]
  126 months (n=14) | 9.00 [1.50 to 60.00]

5. Secondary Outcome: Insulin Antibodies (Percent Binding) by Time on Exubera Treatment - Subjects With Type 2 Diabetes (Using Insulin at Study Entry)
Description: observed values by duration of treatment.
Time Frame: 36 to 126 months
Population: as for outcome 1
Measure: Median (Full Range); unit: percent binding
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 48
percent binding
  36 months (n=22) | 2.75 (14.89) [1.50 to 69.00]
  42 months (n=9) | 1.50 (12.69) [1.50 to 40.00]
  48 months (n=21) | 1.50 [1.50 to 62.00]
  54 months (n=20) | 1.50 [1.50 to 45.00]
  60 months (n=17) | 1.50 [1.50 to 82.00]
  66 months (n=16) | 1.50 [1.50 to 75.00]
  72 months (n=14) | 1.50 [1.50 to 84.00]
  78 months (n=14) | 1.50 [1.50 to 61.00]
  84 months (n=14) | 1.50 [1.50 to 69.00]
  90 months (n=12) | 1.50 [1.50 to 65.00]
  96 months (n=12) | 1.50 [1.50 to 55.00]
  102 months (n=11) | 1.50 [1.50 to 56.00]
  108 months (n=11) | 4.00 [1.50 to 46.00]
  114 months (n=11) | 4.00 [1.50 to 33.00]
  120 months (n=10) | 1.50 [1.50 to 32.00]
  126 months (n=8) | 1.50 [1.50 to 27.00]

6. Primary Outcome: Change in Forced Expiratory Volume in 1 Second (L) by Time on Exubera Treatment
Description: Change from Baseline: mean of (value of observed forced expiratory volume in 1 second (FEV1) (liters) at treatment duration minus baseline value). Duration of treatment is based on the elapsed duration of treatment in the controlled and uncontrolled studies. Baseline was based on pre-inhaled insulin measurements.
Time Frame: Baseline to 126 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 156
liters
  3 months (n=154) | -0.077 (0.204)
  6 months (n=149) | -0.101 (0.204)
  12 months (n=138) | -0.137 (0.220)
  18 months (n=123) | -0.141 (0.218)
  24 months (n=116) | -0.184 (0.232)
  30 months (n=108) | -0.210 (0.237)
  36 months (n=101) | -0.253 (0.244)
  42 months (n=92) | -0.288 (0.217)
  48 months (n=88) | -0.307 (0.252)
  54 months (n=83) | -0.291 (0.260)
  60 months (n=75) | -0.312 (0.267)
  66 months (n=70) | -0.344 (0.273)
  72 months (n=67) | -0.363 (0.289)
  78 months (n=61) | -0.376 (0.281)
  84 months (n=57) | -0.421 (0.301)
  90 months (n=56) | -0.446 (0.311)
  96 months (n=54) | -0.455 (0.332)
  102 months (n=50) | -0.469 (0.321)
  108 months (n=42) | -0.496 (0.273)
  114 months (n=35) | -0.510 (0.281)
  120 months (n=23) | -0.490 (0.298)
  126 months (n=11) | -0.634 (0.371)

7. Secondary Outcome: Insulin Antibodies (Percent Binding) by Time on Exubera Treatment - Subjects With Type 2 Diabetes (Not Using Insulin at Study Entry)
Description: Observed values by duration of treatment.
Time Frame: 6 to 120 months
Population: as for outcome 1
Measure: Median (Full Range); unit: percent binding
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 57
percent binding
  6 months (n=58) | 1.50 (5.36) [1.50 to 29.00]
  12 months (n=48) | 2.25 [1.50 to 55.00]
  18 months (n=5) | 10.00 [1.50 to 19.00]
  24 months (n=41) | 1.50 [1.50 to 44.00]
  30 months (n=4) | 7.25 [1.50 to 28.00]
  36 months (n=37) | 1.50 [1.50 to 41.00]
  42 months (n=33) | 1.50 [1.50 to 38.00]
  48 months (n=32) | 1.50 [1.50 to 43.00]
  54 months (n=30) | 1.50 [1.50 to 43.00]
  60 months (n=25) | 1.50 [1.50 to 42.00]
  66 months (n=30) | 1.50 [1.50 to 40.00]
  72 months (n=24) | 1.50 [1.50 to 36.00]
  78 months (n=23) | 1.50 [1.50 to 54.00]
  84 months (n=20) | 1.50 [1.50 to 41.00]
  90 months (n=18) | 1.50 [1.50 to 48.00]
  96 months (n=18) | 1.50 [1.50 to 50.00]
  102 months (n=14) | 1.50 [1.50 to 36.00]
  108 months (n=13) | 1.50 [1.50 to 24.00]
  114 months (n=9) | 1.50 [1.50 to 20.00]
  120 months (n=6) | 1.50 [1.50 to 5.00]

8. Secondary Outcome: Number of Decliners in Either Forced Expiratory Volume in 1 Second (L) or Carbon Monoxide Diffusing Capacity (ml/Min/mm Hg), by Duration of Exubera Treatment
Description: Decliners = decline of ≥15% in forced expiratory volume or ≥20% in carbon monoxide diffusing capacity.
Time Frame: 3 to >=108 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 156
participants
  3 months (n=154) | 2
  6 months (n=151) | 19
  12 months (n=138) | 14
  18 months (n=123) | 15
  24 months (n=116) | 26
  30 months (n=108) | 26
  36 months (n=101) | 30
  42 months (n=92) | 30
  48 months (n=88) | 24
  54 months (n=83) | 22
  60 months (n=75) | 28
  66 months (n=70) | 25
  72 months (n=67) | 19
  78 months (n=61) | 21
  84 months (n=57) | 26
  90 months (n=56) | 25
  96 months (n=54) | 21
  102 months (n=50) | 25
  >=108 months (n=42) | 29

9. Secondary Outcome: Number of Decliners in Forced Expiratory Volume in 1 Second (L) by Duration of Exubera Treatment
Description: Decliners at particular timepoint were defined as any decline of ≥15% in forced expiratory volume.
Time Frame: 3 to >=108 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 156
participants
  3 months (n=154) | 2
  6 months (n=149) | 5
  12 months (n=138) | 6
  18 months (n=123) | 5
  24 months (n=116) | 9
  30 months (n=108) | 14
  36 months (n=101) | 18
  42 months (n=92) | 18
  48 months (n=88) | 19
  54 months (n=83) | 14
  60 months (n=75) | 21
  66 months (n=70) | 19
  72 months (n=67) | 17
  78 months (n=61) | 17
  84 months (n=57) | 21
  90 months (n=56) | 24
  96 months (n=54) | 19
  102 months (n=50) | 24
  >=108 months (n=42) | 27

10. Secondary Outcome: Number of Decliners in Carbon Monoxide Diffusing Capacity (ml/Min/mm Hg) by Duration of Exubera Treatment
Description: Decliners at particular timepoint were defined as any decline of ≥20% in carbon monoxide diffusing capacity.
Time Frame: 6 to >=108 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 152
participants
  6 months (n=149) | 16
  12 months (n=130) | 8
  18 months (n=115) | 13
  24 months (n=113) | 21
  30 months (n=100) | 14
  36 months (n=95) | 14
  42 months (n=86) | 13
  48 months (n=82) | 11
  54 months (n=80) | 11
  60 months (n=70) | 10
  66 months (n=64) | 11
  72 months (n=62) | 8
  78 months (n=59) | 11
  84 months (n=57) | 10
  90 months (n=50) | 5
  96 months (n=52) | 4
  102 months (n=42) | 4
  >=108 months (n=41) | 13

11. Primary Outcome: Change in Carbon Monoxide Diffusing Capacity (mL/Min/mm Hg) by Time on Exubera Treatment
Description: Change from Baseline: mean of (value of observed Carbon Monoxide Diffusing Capacity (mL/min/mm Hg) at treatment duration minus baseline value). Duration of treatment is based on the elapsed duration of treatment in the controlled and uncontrolled studies. Baseline was based on pre-inhaled insulin measurements.
Time Frame: baseline to 126 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/mm Hg
Arm/Group | Inhaled Insulin
Number analyzed (Participants) | 152
mL/min/mm Hg
  6 months (n=149) | -1.200 (4.358)
  12 months (n=130) | -1.262 (4.446)
  18 months (n=115) | -1.883 (4.690)
  24 months (n=113) | -2.012 (4.821)
  30 months (n=100) | -1.601 (5.816)
  36 months (n=95) | -2.122 (5.030)
  42 months (n=86) | -2.550 (5.307)
  48 months (n=82) | -1.827 (3.623)
  54 months (n=80) | -2.118 (3.485)
  60 months (n=70) | -2.037 (4.325)
  66 months (n=64) | -2.377 (4.168)
  72 months (n=62) | -1.401 (5.061)
  78 months (n=59) | -1.532 (5.764)
  84 months (n=57) | -1.111 (4.672)
  90 months (n=50) | -0.919 (4.043)
  96 months (n=52) | -0.609 (4.763)
  102 months (n=42) | -1.504 (3.514)
  108 months (n=40) | -2.397 (4.496)
  114 months (n=35) | -2.450 (4.471)
  120 months (n=26) | -2.028 (3.403)
  126 months (n=22) | -2.126 (3.984)

ADVERSE EVENTS:
Arm/Group | Inhaled Insulin
Serious Adverse Events (participants affected / at risk) | 63
Other Adverse Events (participants affected / at risk) | 172
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Inhaled Insulin
Impacted colon (Gastrointestinal disorders) | 1/173
Anemia (Blood and lymphatic system disorders) | 2/173
Acute myocardial infarction (Cardiac disorders) | 3/173
Angina pectoris (Cardiac disorders) | 2/173
Angina unstable (Cardiac disorders) | 1/173
Arteriosclerosis coronary artery (Cardiac disorders) | 1/173
Bradycardia (Cardiac disorders) | 2/173
Cardiac failure congestive (Cardiac disorders) | 3/173
Cardio-respiratory arrest (Cardiac disorders) | 1/173
Coronary artery disease (Cardiac disorders) | 10/173
Coronary artery occlusion (Cardiac disorders) | 2/173
Coronary artery stenosis (Cardiac disorders) | 1/173
Myocardial infarction (Cardiac disorders) | 5/173
Myocardial ischaemia (Cardiac disorders) | 1/173
Tachycardia (Cardiac disorders) | 1/173
Ventricular extrasystoles (Cardiac disorders) | 1/173
Vertigo (Ear and labyrinth disorders) | 1/173
Goitre (Endocrine disorders) | 1/173
Vitreous haemorrhage (Eye disorders) | 1/173
Duodenal ulcer (Gastrointestinal disorders) | 1/173
Food poisoning (Gastrointestinal disorders) | 1/173
Haemorrhagic ascites (Gastrointestinal disorders) | 1/173
Nausea (Gastrointestinal disorders) | 1/173
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/173
Vomiting (Gastrointestinal disorders) | 1/173
Chest pain (General disorders) | 6/173
Impaired healing (General disorders) | 1/173
Non-cardiac chest pain (General disorders) | 1/173
Pain (General disorders) | 1/173
Cholelithiasis (Hepatobiliary disorders) | 2/173
Jaundice (Hepatobiliary disorders) | 1/173
Abdominal wall abscess (Infections and infestations) | 1/173
Bronchitis (Infections and infestations) | 1/173
Cellulitis (Infections and infestations) | 1/173
Cholecystitis infective (Infections and infestations) | 1/173
Diverticulitis (Infections and infestations) | 1/173
Gastroenteritis (Infections and infestations) | 1/173
Localised infection (Infections and infestations) | 1/173
Periorbital cellulitis (Infections and infestations) | 1/173
Pneumonia (Infections and infestations) | 2/173
Pyelonephritis (Infections and infestations) | 1/173
Urosepsis (Infections and infestations) | 1/173
Ankle fracture (Injury, poisoning and procedural complications) | 1/173
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1/173
Clavicle fracture (Injury, poisoning and procedural complications) | 1/173
Foot fracture (Injury, poisoning and procedural complications) | 1/173
Humerus fracture (Injury, poisoning and procedural complications) | 1/173
Laceration (Injury, poisoning and procedural complications) | 1/173
Radius fracture (Injury, poisoning and procedural complications) | 1/173
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1/173
Rib fracture (Injury, poisoning and procedural complications) | 2/173
Road traffic accident (Injury, poisoning and procedural complications) | 4/173
Upper limb fracture (Injury, poisoning and procedural complications) | 1/173
Hepatic enzyme increased (Investigations) | 1/173
Oxygen saturation decreased (Investigations) | 1/173
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1/173
Fluid overload (Metabolism and nutrition disorders) | 1/173
Hyperkalaemia (Metabolism and nutrition disorders) | 1/173
Hypoglycaemia (Metabolism and nutrition disorders) | 1/173
Hypokalaemia (Metabolism and nutrition disorders) | 1/173
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/173
Back pain (Musculoskeletal and connective tissue disorders) | 2/173
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2/173
Spondylitis (Musculoskeletal and connective tissue disorders) | 1/173
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/173
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/173
Central nervous system lympoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Cerebrovascular accident (Nervous system disorders) | 2/173
Haemorrhage intracranial (Nervous system disorders) | 1/173
Loss of consciousness (Nervous system disorders) | 1/173
Paraplegia (Nervous system disorders) | 1/173
Syncope (Nervous system disorders) | 2/173
Transient ischaemic attack (Nervous system disorders) | 1/173
Dysuria (Renal and urinary disorders) | 1/173
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/173
Erectile dysfunction (Reproductive system and breast disorders) | 1/173
Fallopian tube cyst (Reproductive system and breast disorders) | 1/173
Fallopian tube disorder (Reproductive system and breast disorders) | 1/173
Menorrhagia (Reproductive system and breast disorders) | 1/173
Ovarian cyst (Reproductive system and breast disorders) | 2/173
Pelvic peritoneal adhesions (Reproductive system and breast disorders) | 1/173
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/173
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1/173
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/173
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/173
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/173
Cardiac pacemaker insertion (Surgical and medical procedures) | 1/173
Aortic stenosis (Vascular disorders) | 1/173
Arterial thrombosis (Vascular disorders) | 1/173
Arterial thrombosis limb (Vascular disorders) | 1/173
Thrombosis (Vascular disorders) | 1/173
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Inhaled Insulin
Anaemia (Blood and lymphatic system disorders) | 7/173
Lymphadenitis (Blood and lymphatic system disorders) | 1/173
Lymphadenopathy (Blood and lymphatic system disorders) | 5/173
Acute myocardial infarction (Cardiac disorders) | 3/173
Angina pectoris (Cardiac disorders) | 4/173
Angina unstable (Cardiac disorders) | 1/173
Arteriosclerosis coronary artery (Cardiac disorders) | 1/173
Bradycardia (Cardiac disorders) | 2/173
Bundle branch block right (Cardiac disorders) | 1/173
Cardiac aneurysm (Cardiac disorders) | 1/173
Cardiac failure congestive (Cardiac disorders) | 3/173
Cardio-respiratory arrest (Cardiac disorders) | 1/173
Cardiomegaly (Cardiac disorders) | 4/173
Coronary artery disease (Cardiac disorders) | 14/173
Coronary artery occlusion (Cardiac disorders) | 2/173
Coronary artery stenosis (Cardiac disorders) | 1/173
Left atrial dilatation (Cardiac disorders) | 1/173
Myocardial infarction (Cardiac disorders) | 5/173
Myocardial ischaemia (Cardiac disorders) | 1/173
Palpitations (Cardiac disorders) | 11/173
Sinus arrhythmia (Cardiac disorders) | 1/173
Sinus tachycardia (Cardiac disorders) | 1/173
Supraventricular extrasystoles (Cardiac disorders) | 1/173
Supraventricular tachycardia (Cardiac disorders) | 1/173
Tachycardia (Cardiac disorders) | 6/173
Ventricular extrasystoles (Cardiac disorders) | 2/173
Familial tremor (Congenital, familial and genetic disorders) | 1/173
Auricular swelling (Ear and labyrinth disorders) | 1/173
Cerumen impaction (Ear and labyrinth disorders) | 1/173
Deafness (Ear and labyrinth disorders) | 1/173
Deafness unilateral (Ear and labyrinth disorders) | 1/173
Ear canal erythema (Ear and labyrinth disorders) | 1/173
Ear congestion (Ear and labyrinth disorders) | 1/173
Ear discomfort (Ear and labyrinth disorders) | 7/173
Ear disorder (Ear and labyrinth disorders) | 3/173
Ear pain (Ear and labyrinth disorders) | 12/173
Eustachian tube dysfunction (Ear and labyrinth disorders) | 2/173
Hypoacusis (Ear and labyrinth disorders) | 2/173
Meniere's disease (Ear and labyrinth disorders) | 3/173
Motion sickness (Ear and labyrinth disorders) | 1/173
Otorrhoea (Ear and labyrinth disorders) | 2/173
Tinnitus (Ear and labyrinth disorders) | 4/173
Tympanic membrane disorder (Ear and labyrinth disorders) | 1/173
Tympanic membrane perforation (Ear and labyrinth disorders) | 1/173
Vertigo (Ear and labyrinth disorders) | 7/173
Androgen deficiency (Endocrine disorders) | 1/173
Goitre (Endocrine disorders) | 3/173
Hypothyroidism (Endocrine disorders) | 5/173
Thyroid pain (Endocrine disorders) | 1/173
Cataract (Eye disorders) | 9/173
Cataract nuclear (Eye disorders) | 2/173
Conjunctival haemorrhage (Eye disorders) | 1/173
Conjunctivitis (Eye disorders) | 4/173
Diabetic retinopathy (Eye disorders) | 15/173
Diplopia (Eye disorders) | 2/173
Dry eye (Eye disorders) | 2/173
Eye allergy (Eye disorders) | 1/173
Eye discharge (Eye disorders) | 2/173
Eye haemorrhage (Eye disorders) | 3/173
Eye inflammation (Eye disorders) | 1/173
Eye irritation (Eye disorders) | 2/173
Eye movement disorder (Eye disorders) | 2/173
Eye pain (Eye disorders) | 1/173
Glaucoma (Eye disorders) | 4/173
Hyphaema (Eye disorders) | 1/173
Iridocyclitis (Eye disorders) | 1/173
Lacrimation increased (Eye disorders) | 2/173
Macular degeneration (Eye disorders) | 1/173
Macular oedema (Eye disorders) | 2/173
Myodesopsia (Eye disorders) | 2/173
Photopsia (Eye disorders) | 2/173
Retinal aneurysm (Eye disorders) | 2/173
Retinal detachment (Eye disorders) | 1/173
Retinal haemorrhage (Eye disorders) | 1/173
Retinopathy (Eye disorders) | 6/173
Scotoma (Eye disorders) | 1/173
Vision blurred (Eye disorders) | 20/173
Visual acuity reduced (Eye disorders) | 1/173
Visual impairment (Eye disorders) | 2/173
Vitreous haemorrhage (Eye disorders) | 2/173
Abdominal discomfort (Gastrointestinal disorders) | 9/173
Abdominal distension (Gastrointestinal disorders) | 2/173
Abdominal pain (Gastrointestinal disorders) | 19/173
Abdominal pain lower (Gastrointestinal disorders) | 5/173
Abdominal pain upper (Gastrointestinal disorders) | 19/173
Breath odour (Gastrointestinal disorders) | 1/173
Colitis (Gastrointestinal disorders) | 1/173
Colonic Polyp (Gastrointestinal disorders) | 3/173
Constipation (Gastrointestinal disorders) | 18/173
Dental caries (Gastrointestinal disorders) | 6/173
Diarrhoea (Gastrointestinal disorders) | 45/173
Diverticulum (Gastrointestinal disorders) | 3/173
Dry mouth (Gastrointestinal disorders) | 5/173
Duodenal ulcer (Gastrointestinal disorders) | 1/173
Duodenogastric reflux (Gastrointestinal disorders) | 2/173
Dyspepsia (Gastrointestinal disorders) | 21/173
Dysphagia (Gastrointestinal disorders) | 2/173
Faecal incontinence (Gastrointestinal disorders) | 1/173
Faeces discoloured (Gastrointestinal disorders) | 1/173
Flatulence (Gastrointestinal disorders) | 2/173
Food poisoning (Gastrointestinal disorders) | 6/173
Frequent bowel movements (Gastrointestinal disorders) | 1/173
Gastric ulcer (Gastrointestinal disorders) | 1/173
Gastritis (Gastrointestinal disorders) | 2/173
Gastrointestinal pain (Gastrointestinal disorders) | 1/173
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 17/173
Gingival pain (Gastrointestinal disorders) | 3/173
Gingival recession (Gastrointestinal disorders) | 1/173
Gingival swelling (Gastrointestinal disorders) | 1/173
Gingivitis (Gastrointestinal disorders) | 3/173
Glossitis (Gastrointestinal disorders) | 1/173
Haematochezia (Gastrointestinal disorders) | 1/173
Haemorrhagic ascites (Gastrointestinal disorders) | 1/173
Haemorrhoids (Gastrointestinal disorders) | 7/173
Hiatus hernia (Gastrointestinal disorders) | 2/173
Hypoaesthesia oral (Gastrointestinal disorders) | 4/173
Impaired gastric emptying (Gastrointestinal disorders) | 3/173
Inguinal hernia (Gastrointestinal disorders) | 1/173
Irritable bowel syndrome (Gastrointestinal disorders) | 1/173
Lip blister (Gastrointestinal disorders) | 2/173
Lip disorder (Gastrointestinal disorders) | 1/173
Mouth ulceration (Gastrointestinal disorders) | 1/173
Nausea (Gastrointestinal disorders) | 48/173
Paraesthesia oral (Gastrointestinal disorders) | 4/173
Parotid gland enlargement (Gastrointestinal disorders) | 1/173
Periodontal disease (Gastrointestinal disorders) | 3/173
Rectal haemorrhage (Gastrointestinal disorders) | 1/173
Rectal polyp (Gastrointestinal disorders) | 2/173
Reflux oesophagitis (Gastrointestinal disorders) | 1/173
Retching (Gastrointestinal disorders) | 2/173
Stomach discomfort (Gastrointestinal disorders) | 7/173
Swollen tongue (Gastrointestinal disorders) | 1/173
Tongue discolouration (Gastrointestinal disorders) | 2/173
Tongue disorder (Gastrointestinal disorders) | 2/173
Tooth impacted (Gastrointestinal disorders) | 1/173
Tooth loss (Gastrointestinal disorders) | 1/173
Toothache (Gastrointestinal disorders) | 18/173
Umbilical hernia (Gastrointestinal disorders) | 2/173
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/173
Vomiting (Gastrointestinal disorders) | 24/173
Asthenia (General disorders) | 41/173
Catheter site inflammation (General disorders) | 1/173
Chest discomfort (General disorders) | 5/173
Chest pain (General disorders) | 23/173
Chills (General disorders) | 3/173
Cyst (General disorders) | 2/173
Discomfort (General disorders) | 1/173
Face oedema (General disorders) | 2/173
Fatigue (General disorders) | 38/173
Feeling abnormal (General disorders) | 3/173
Feeling cold (General disorders) | 3/173
Feeling hot (General disorders) | 3/173
Feeling jittery (General disorders) | 9/173
Generalised oedema (General disorders) | 7/173
Hunger (General disorders) | 24/173
Ill-defined disorder (General disorders) | 1/173
Impaired healing (General disorders) | 1/173
Influenza like illness (General disorders) | 3/173
Injection site pain (General disorders) | 1/173
Injection site pruritus (General disorders) | 1/173
Irritability (General disorders) | 5/173
Malaise (General disorders) | 8/173
Non-cardiac chest pain (General disorders) | 1/173
Oedema (General disorders) | 3/173
Oedema peripheral (General disorders) | 34/173
Pain (General disorders) | 14/173
Peripheral coldness (General disorders) | 1/173
Pitting oedema (General disorders) | 1/173
Pyrexia (General disorders) | 12/173
Sensation of foreign body (General disorders) | 2/173
Sluggishness (General disorders) | 3/173
Temperature intolerance (General disorders) | 1/173
Thirst (General disorders) | 4/173
Cholelithiasis (Hepatobiliary disorders) | 3/173
Hepatic steatosis (Hepatobiliary disorders) | 2/173
Jaundice (Hepatobiliary disorders) | 1/173
Liver disorder (Hepatobiliary disorders) | 1/173
Anaphylactic reaction (Immune system disorders) | 1/173
Drug hypersensitivity (Immune system disorders) | 1/173
Hypersensitivity (Immune system disorders) | 8/173
Latex allergy (Immune system disorders) | 1/173
Seasonal allergy (Immune system disorders) | 20/173
Abdominal wall abscess (Infections and infestations) | 1/173
Abscess limb (Infections and infestations) | 2/173
Acarodermatitis (Infections and infestations) | 1/173
Acute sinusitis (Infections and infestations) | 1/173
Breast abscess (Infections and infestations) | 1/173
Bronchitis (Infections and infestations) | 30/173
Candidiasis (Infections and infestations) | 1/173
Catheter related infection (Infections and infestations) | 1/173
Catheter site infection (Infections and infestations) | 1/173
Cellulitis (Infections and infestations) | 7/173
Cholecystitis infective (Infections and infestations) | 1/173
Chronic sinusitis (Infections and infestations) | 1/173
Conjunctivitis infective (Infections and infestations) | 1/173
Cystitis (Infections and infestations) | 5/173
Diverticulitis (Infections and infestations) | 2/173
Ear infection (Infections and infestations) | 3/173
Erythema infectiosum (Infections and infestations) | 1/173
Eye infection (Infections and infestations) | 1/173
Folliculitis (Infections and infestations) | 2/173
Fungal infection (Infections and infestations) | 6/173
Fungal skin infection (Infections and infestations) | 4/173
Furuncle (Infections and infestations) | 7/173
Gastric infection (Infections and infestations) | 1/173
Gastroenteritis (Infections and infestations) | 16/173
Gastroenteritis viral (Infections and infestations) | 32/173
Genital infection fungal (Infections and infestations) | 1/173
Groin Abscess (Infections and infestations) | 1/173
Herpes simplex (Infections and infestations) | 1/173
Herpes zosters (Infections and infestations) | 7/173
Hordeolum (Infections and infestations) | 3/173
Infected cyst (Infections and infestations) | 1/173
Infected sebaceous cyst (Infections and infestations) | 2/173
Infected skin ulcer (Infections and infestations) | 1/173
Infection (Infections and infestations) | 4/173
Infectious mononucleosis (Infections and infestations) | 1/173
Influenza (Infections and infestations) | 50/173
Kidney infection (Infections and infestations) | 2/173
Labyrinthitis (Infections and infestations) | 4/173
Laryngitis (Infections and infestations) | 7/173
Localised infection (Infections and infestations) | 10/173
Lower respiratory tract infection (Infections and infestations) | 6/173
Lymph gland infection (Infections and infestations) | 1/173
Gingival infection (Infections and infestations) | 5/173
Nail bed infection (Infections and infestations) | 2/173
Nasopharyngitis (Infections and infestations) | 34/173
Onychomycosis (Infections and infestations) | 11/173
Oral herpes (Infections and infestations) | 6/173
Osteomyelitis (Infections and infestations) | 1/173
Otitis externa (Infections and infestations) | 5/173
Otitis media (Infections and infestations) | 11/173
Paronychia (Infections and infestations) | 2/173
Penile infection (Infections and infestations) | 1/173
Periorbital cellulitis (Infections and infestations) | 1/173
Pharyngitis (Infections and infestations) | 17/173
Pharyngitis streptococcal (Infections and infestations) | 9/173
Pneumonia (Infections and infestations) | 10/173
Postoperative wound infection (Infections and infestations) | 2/173
Pyelonephritis (Infections and infestations) | 2/173
Recurring skin boils (Infections and infestations) | 1/173
Respiratory tract infection (Infections and infestations) | 1/173
Rhinitis (Infections and infestations) | 7/173
Scrotal abscess (Infections and infestations) | 1/173
Sinusitis (Infections and infestations) | 33/173
Skin infection (Infections and infestations) | 1/173
Soft tissue infection (Infections and infestations) | 1/173
Subcutaneous abscess (Infections and infestations) | 1/173
Tinea infection (Infections and infestations) | 1/173
Tinea pedis (Infections and infestations) | 6/173
Tonsillitis (Infections and infestations) | 2/173
Tooth abscess (Infections and infestations) | 10/173
Tooth infection (Infections and infestations) | 8/173
Upper respiratory tract infection (Infections and infestations) | 102/173
Urinary tract infection (Infections and infestations) | 26/173
Urosepsis (Infections and infestations) | 1/173
Vaginal infection (Infections and infestations) | 4/173
Vaginitis bacterial (Infections and infestations) | 1/173
Viral infection (Infections and infestations) | 9/173
Viral pharyngitis (Infections and infestations) | 1/173
Viral upper respiratory tract infection (Infections and infestations) | 1/173
Vulval abscess (Infections and infestations) | 1/173
Vulvovaginal mycotic infection (Infections and infestations) | 13/173
Wound infection (Infections and infestations) | 3/173
Animal bite (Injury, poisoning and procedural complications) | 1/173
Ankle fracture (Injury, poisoning and procedural complications) | 3/173
Arthropod bite (Injury, poisoning and procedural complications) | 1/173
Arthropod sting (Injury, poisoning and procedural complications) | 1/173
Back injury (Injury, poisoning and procedural complications) | 6/173
Barotitis media (Injury, poisoning and procedural complications) | 1/173
Burns second degree (Injury, poisoning and procedural complications) | 2/173
Burns third degree (Injury, poisoning and procedural complications) | 1/173
Cartilage injury (Injury, poisoning and procedural complications) | 3/173
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2/173
Clavicle fracture (Injury, poisoning and procedural complications) | 2/173
Contusion (Injury, poisoning and procedural complications) | 16/173
Device failure (Injury, poisoning and procedural complications) | 1/173
Epicondylitis (Injury, poisoning and procedural complications) | 3/173
Excoriation (Injury, poisoning and procedural complications) | 19/173
Eye injury (Injury, poisoning and procedural complications) | 1/173
Foot fracture (Injury, poisoning and procedural complications) | 11/173
Hand fracture (Injury, poisoning and procedural complications) | 4/173
Humerus fracture (Injury, poisoning and procedural complications) | 1/173
Incision site pain (Injury, poisoning and procedural complications) | 3/173
Injury (Injury, poisoning and procedural complications) | 1/173
Injury corneal (Injury, poisoning and procedural complications) | 1/173
Joint dislocation (Injury, poisoning and procedural complications) | 1/173
Joint injury (Injury, poisoning and procedural complications) | 2/173
Joint sprain (Injury, poisoning and procedural complications) | 11/173
Laceration (Injury, poisoning and procedural complications) | 9/173
Ligament rupture (Injury, poisoning and procedural complications) | 1/173
Limb injury (Injury, poisoning and procedural complications) | 2/173
Lung injury (Injury, poisoning and procedural complications) | 1/173
Meniscus lesion (Injury, poisoning and procedural complications) | 2/173
Muscle injury (Injury, poisoning and procedural complications) | 3/173
Muscle strain (Injury, poisoning and procedural complications) | 12/173
Open fracture (Injury, poisoning and procedural complications) | 1/173
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1/173
Procedural pain (Injury, poisoning and procedural complications) | 8/173
Radius fracture (Injury, poisoning and procedural complications) | 1/173
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1/173
Rib fracture (Injury, poisoning and procedural complications) | 6/173
Road traffic accident (Injury, poisoning and procedural complications) | 5/173
Skeletal injury (Injury, poisoning and procedural complications) | 6/173
Skin laceration (Injury, poisoning and procedural complications) | 8/173
Stress fracture (Injury, poisoning and procedural complications) | 1/173
Sunburn (Injury, poisoning and procedural complications) | 1/173
Tendon injury (Injury, poisoning and procedural complications) | 2/173
Tendon rupture (Injury, poisoning and procedural complications) | 1/173
Thermal burn (Injury, poisoning and procedural complications) | 8/173
Tooth fracture (Injury, poisoning and procedural complications) | 3/173
Upper limb fracture (Injury, poisoning and procedural complications) | 1/173
Wound (Injury, poisoning and procedural complications) | 3/173
Wrist fracture (Injury, poisoning and procedural complications) | 1/173
Aspartate aminotransferase increased (Investigations) | 2/173
Blood cholesterol increased (Investigations) | 1/173
Blood pressure increased (Investigations) | 5/173
Blood testosterone decreased (Investigations) | 2/173
Blood urine present (Investigations) | 1/173
Bone density decreased (Investigations) | 1/173
Cardiac murmur (Investigations) | 1/173
Cardiac stress test abnormal (Investigations) | 1/173
Carotid bruit (Investigations) | 1/173
Chest X-ray abnormal (Investigations) | 1/173
Culture (Investigations) | 1/173
Full blood count decreased (Investigations) | 1/173
Glycosylated haemoglobin (Investigations) | 1/173
Heart rate increased (Investigations) | 6/173
Heart rate irregular (Investigations) | 2/173
Hepatic enzyme increased (Investigations) | 1/173
Occult blood positive (Investigations) | 2/173
Oxygen saturation decreased (Investigations) | 1/173
Platelet count decreased (Investigations) | 2/173
Pulmonary function test decreased (Investigations) | 2/173
Pulse abnormal (Investigations) | 1/173
Smear cervix abnormal (Investigations) | 1/173
Urine analysis abnormal (Investigations) | 1/173
Vitamin B12 decreased (Investigations) | 1/173
Weight increased (Investigations) | 2/173
White blood cell count decreased (Investigations) | 1/173
Anorexia (Metabolism and nutrition disorders) | 1/173
Dehydration (Metabolism and nutrition disorders) | 1/173
Diabetic foot (Metabolism and nutrition disorders) | 2/173
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1/173
Dyslipidaemia (Metabolism and nutrition disorders) | 1/173
Fluid overload (Metabolism and nutrition disorders) | 1/173
Fluid retention (Metabolism and nutrition disorders) | 2/173
Hypercalcaemia (Metabolism and nutrition disorders) | 1/173
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5/173
Hyperglycaemia (Metabolism and nutrition disorders) | 6/173
Hyperkalaemia (Metabolism and nutrition disorders) | 2/173
Hyperlipidaemia (Metabolism and nutrition disorders) | 7/173
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1/173
Hypoglycaemia (Metabolism and nutrition disorders) | 125/173
Hypokalaemia (Metabolism and nutrition disorders) | 4/173
Ketosis (Metabolism and nutrition disorders) | 1/173
Lactic acidosis (Metabolism and nutrition disorders) | 1/173
Polydipsia (Metabolism and nutrition disorders) | 2/173
Arthralgia (Musculoskeletal and connective tissue disorders) | 52/173
Arthritis (Musculoskeletal and connective tissue disorders) | 6/173
Arthropathy (Musculoskeletal and connective tissue disorders) | 3/173
Back pain (Musculoskeletal and connective tissue disorders) | 42/173
Bone pain (Musculoskeletal and connective tissue disorders) | 2/173
Bursitis (Musculoskeletal and connective tissue disorders) | 5/173
Coccydynia (Musculoskeletal and connective tissue disorders) | 1/173
Costochondritis (Musculoskeletal and connective tissue disorders) | 1/173
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2/173
Exostosis (Musculoskeletal and connective tissue disorders) | 7/173
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1/173
Flank pain (Musculoskeletal and connective tissue disorders) | 2/173
Foot deformity (Musculoskeletal and connective tissue disorders) | 2/173
Groin pain (Musculoskeletal and connective tissue disorders) | 1/173
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1/173
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6/173
Joint contracture (Musculoskeletal and connective tissue disorders) | 1/173
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3/173
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3/173
Joint swelling (Musculoskeletal and connective tissue disorders) | 4/173
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2/173
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/173
Monarthritis (Musculoskeletal and connective tissue disorders) | 1/173
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1/173
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18/173
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1/173
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3/173
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14/173
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 4/173
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2/173
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23/173
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4/173
Myalgia (Musculoskeletal and connective tissue disorders) | 11/173
Neck pain (Musculoskeletal and connective tissue disorders) | 8/173
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1/173
Osteitis (Musculoskeletal and connective tissue disorders) | 1/173
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4/173
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1/173
Osteopenia (Musculoskeletal and connective tissue disorders) | 2/173
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48/173
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2/173
Periarthritis (Musculoskeletal and connective tissue disorders) | 2/173
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1/173
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1/173
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2/173
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1/173
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1/173
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/173
Spondylitis (Musculoskeletal and connective tissue disorders) | 2/173
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1/173
Synovitis (Musculoskeletal and connective tissue disorders) | 1/173
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1/173
Tendonitis (Musculoskeletal and connective tissue disorders) | 19/173
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2/173
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1/173
Trigger finger (Musculoskeletal and connective tissue disorders) | 5/173
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 1/173
CARPAL TUNNEL SYNDROME - RIGHT WRIST (Nervous system disorders) | 1/173
DECREASED BREATHING BILATERALLY (Respiratory, thoracic and mediastinal disorders) | 1/173
DRY, PEELING LIPS (Gastrointestinal disorders) | 1/173
IMPACTED COLON (Gastrointestinal disorders) | 1/173
LIGHT SENSITIVE VISION (Eye disorders) | 1/173
PROGRESSION OF PROLIFERATIVE DIABETIC RETINOPATHY OF LEFT EYE (Eye disorders) | 1/173
PROGRESSION OF PROLIFERATIVE DIABETIC RETINOPATHY RIGHT EYE (Eye disorders) | 1/173
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/173
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/173
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/173
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/173
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/173
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/173
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/173
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/173
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/173
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/173
Areflexia (Nervous system disorders) | 1/173
Burning sensation (Nervous system disorders) | 4/173
Carpal tunnel syndrome (Nervous system disorders) | 10/173
Cerebrovascular accident (Nervous system disorders) | 2/173
Cognitive disorder (Nervous system disorders) | 1/173
Coordination abnormal (Nervous system disorders) | 1/173
Diabetic neuropathy (Nervous system disorders) | 2/173
Disturbance in attention (Nervous system disorders) | 5/173
Dizziness (Nervous system disorders) | 46/173
Dizziness postural (Nervous system disorders) | 1/173
Dysgeusia (Nervous system disorders) | 1/173
Facial palsy (Nervous system disorders) | 2/173
Haemorrhage intracranial (Nervous system disorders) | 1/173
Head discomfort (Nervous system disorders) | 1/173
Headache (Nervous system disorders) | 45/173
Hyperaesthesia (Nervous system disorders) | 1/173
Hypoaesthesia (Nervous system disorders) | 26/173
IIIrd nerve paralysis (Nervous system disorders) | 1/173
Lethargy (Nervous system disorders) | 9/173
Loss of consciousness (Nervous system disorders) | 2/173
Lumbar radiculopathy (Nervous system disorders) | 1/173
Memory impairment (Nervous system disorders) | 3/173
Mental impairment (Nervous system disorders) | 2/173
Migraine (Nervous system disorders) | 4/173
Morton's neuralgia (Nervous system disorders) | 1/173
Nerve compression (Nervous system disorders) | 3/173
Neuralgia (Nervous system disorders) | 3/173
Paraesthesia (Nervous system disorders) | 20/173
Paraplegia (Nervous system disorders) | 1/173
Parkinson's disease (Nervous system disorders) | 1/173
Polyneuropathy (Nervous system disorders) | 1/173
Poor quality sleep (Nervous system disorders) | 1/173
Sciatic nerve neuropathy (Nervous system disorders) | 1/173
Sciatica (Nervous system disorders) | 5/173
Sinus headache (Nervous system disorders) | 11/173
Speech disorder (Nervous system disorders) | 1/173
Syncope (Nervous system disorders) | 5/173
Tension headache (Nervous system disorders) | 2/173
Tinel's sign (Nervous system disorders) | 1/173
Transient ischaemic attack (Nervous system disorders) | 2/173
Tremor (Nervous system disorders) | 62/173
VIth nerve paralysis (Nervous system disorders) | 1/173
Abnormal dreams (Psychiatric disorders) | 1/173
Agitation (Psychiatric disorders) | 2/173
Anxiety (Nervous system disorders) | 23/173
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1/173
Bipolar disorder (Psychiatric disorders) | 1/173
Confusional state (Psychiatric disorders) | 7/173
Daydreaming (Psychiatric disorders) | 1/173
Depression (Psychiatric disorders) | 20/173
Disorientation (Psychiatric disorders) | 9/173
Dissociation (Psychiatric disorders) | 1/173
Emotional disorder (Psychiatric disorders) | 3/173
Flat affect (Psychiatric disorders) | 1/173
Intentional self-injury (Nervous system disorders) | 1/173
Mental status changes (Psychiatric disorders) | 1/173
Mood altered (Psychiatric disorders) | 1/173
Nervousness (Psychiatric disorders) | 17/173
Nightmare (Psychiatric disorders) | 1/173
Restlessness (Psychiatric disorders) | 3/173
Sleep disorder (Psychiatric disorders) | 4/173
Stress (Psychiatric disorders) | 20/173
Thinking abnormal (Psychiatric disorders) | 1/173
Bladder spasm (Renal and urinary disorders) | 1/173
Dysuria (Renal and urinary disorders) | 5/173
Haematuria (Renal and urinary disorders) | 3/173
Hydronephrosis (Renal and urinary disorders) | 1/173
Hypercalciuria (Renal and urinary disorders) | 1/173
Microalbuminuria (Renal and urinary disorders) | 7/173
Micturition disorder (Renal and urinary disorders) | 1/173
Micturition urgency (Renal and urinary disorders) | 3/173
Nephrolithiasis (Renal and urinary disorders) | 7/173
Nephropathy (Renal and urinary disorders) | 2/173
Nephrotic syndrome (Renal and urinary disorders) | 1/173
Nocturia (Renal and urinary disorders) | 2/173
Pollakiuria (Renal and urinary disorders) | 5/173
Polyuria (Renal and urinary disorders) | 5/173
Proteinuria (Renal and urinary disorders) | 3/173
Renal cyst (Renal and urinary disorders) | 1/173
Renal failure (Renal and urinary disorders) | 1/173
Renal failure chronic (Renal and urinary disorders) | 1/173
Stress urinary incontinence (Renal and urinary disorders) | 2/173
Urinary incontinence (Renal and urinary disorders) | 2/173
Urinary tract obstruction (Renal and urinary disorders) | 1/173
Urine odour abnormal (Renal and urinary disorders) | 1/173
Amenorrhoea (Reproductive system and breast disorders) | 2/173
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1/173
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/173
Breast mass (Reproductive system and breast disorders) | 1/173
Breast pain (Reproductive system and breast disorders) | 1/173
Breast tenderness (Reproductive system and breast disorders) | 1/173
Cervical polyp (Reproductive system and breast disorders) | 1/173
Dysmenorrhoea (Reproductive system and breast disorders) | 3/173
Erectile dysfunction (Reproductive system and breast disorders) | 14/173
Fallopian tube cyst (Reproductive system and breast disorders) | 1/173
Fallopian tube disorder (Reproductive system and breast disorders) | 1/173
Menorrhagia (Reproductive system and breast disorders) | 3/173
Menstruation irregular (Reproductive system and breast disorders) | 2/173
Ovarian cyst (Reproductive system and breast disorders) | 2/173
Pelvic peritoneal adhesions (Reproductive system and breast disorders) | 1/173
Peyronie's disease (Reproductive system and breast disorders) | 1/173
Prostatomegaly (Reproductive system and breast disorders) | 2/173
Testicular cyst (Reproductive system and breast disorders) | 1/173
Testicular pain (Reproductive system and breast disorders) | 1/173
Uterine haemorrhage (Reproductive system and breast disorders) | 1/173
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/173
Vulva cyst (Reproductive system and breast disorders) | 1/173
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/173
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1/173
Asthma (Respiratory, thoracic and mediastinal disorders) | 7/173
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1/173
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2/173
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 1/173
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/173
Cough (Respiratory, thoracic and mediastinal disorders) | 70/173
Dry throat (Respiratory, thoracic and mediastinal disorders) | 4/173
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4/173
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16/173
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4/173
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4/173
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1/173
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1/173
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1/173
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3/173
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1/173
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23/173
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1/173
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1/173
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2/173
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 40/173
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1/173
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2/173
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/173
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/173
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1/173
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1/173
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/173
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 9/173
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12/173
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 10/173
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/173
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1/173
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1/173
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/173
Rales (Respiratory, thoracic and mediastinal disorders) | 4/173
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2/173
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/173
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 2/173
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1/173
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1/173
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1/173
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 18/173
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 2/173
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9/173
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 31/173
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1/173
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 7/173
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1/173
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 10/173
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1/173
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7/173
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7/173
Acrodermatitis (Skin and subcutaneous tissue disorders) | 4/173
Alopecia (Skin and subcutaneous tissue disorders) | 2/173
Blister (Skin and subcutaneous tissue disorders) | 6/173
Cold sweat (Skin and subcutaneous tissue disorders) | 6/173
Dandruff (Skin and subcutaneous tissue disorders) | 1/173
Dermal cyst (Skin and subcutaneous tissue disorders) | 6/173
Dermatitis (Skin and subcutaneous tissue disorders) | 5/173
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1/173
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2/173
Dry skin (Skin and subcutaneous tissue disorders) | 7/173
Ecchymosis (Skin and subcutaneous tissue disorders) | 1/173
Eczema (Skin and subcutaneous tissue disorders) | 2/173
Erythema (Skin and subcutaneous tissue disorders) | 3/173
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1/173
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 34/173
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 6/173
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 2/173
Ingrowing nail (Skin and subcutaneous tissue disorders) | 9/173
Nail discomfort (Skin and subcutaneous tissue disorders) | 1/173
Nail disorder (Skin and subcutaneous tissue disorders) | 1/173
Night sweats (Skin and subcutaneous tissue disorders) | 2/173
Onychoclasis (Skin and subcutaneous tissue disorders) | 1/173
Onychogryphosis (Skin and subcutaneous tissue disorders) | 1/173
Onychomadesis (Skin and subcutaneous tissue disorders) | 1/173
Pain of skin (Skin and subcutaneous tissue disorders) | 1/173
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1/173
Pruritus (Skin and subcutaneous tissue disorders) | 3/173
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2/173
Psoriasis (Skin and subcutaneous tissue disorders) | 2/173
Purpura (Skin and subcutaneous tissue disorders) | 1/173
Rash (Skin and subcutaneous tissue disorders) | 24/173
Rash generalised (Skin and subcutaneous tissue disorders) | 3/173
Rash macular (Skin and subcutaneous tissue disorders) | 3/173
Rash papular (Skin and subcutaneous tissue disorders) | 3/173
Rash pruritic (Skin and subcutaneous tissue disorders) | 1/173
Rash vesicular (Skin and subcutaneous tissue disorders) | 1/173
Rosacea (Skin and subcutaneous tissue disorders) | 2/173
Seborrhoea (Skin and subcutaneous tissue disorders) | 1/173
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1/173
Skin discolouration (Skin and subcutaneous tissue disorders) | 3/173
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2/173
Skin irritation (Skin and subcutaneous tissue disorders) | 3/173
Skin lesion (Skin and subcutaneous tissue disorders) | 9/173
Skin nodule (Skin and subcutaneous tissue disorders) | 2/173
Skin ulcer (Skin and subcutaneous tissue disorders) | 10/173
Swelling face (Skin and subcutaneous tissue disorders) | 1/173
Urticaria (Skin and subcutaneous tissue disorders) | 6/173
Family stress (Social circumstances) | 2/173
Menopause (Social circumstances) | 1/173
Cardiac pacemaker insertion (Surgical and medical procedures) | 1/173
Female sterilisation (Surgical and medical procedures) | 1/173
Prophylaxis (Surgical and medical procedures) | 1/173
Sebaceous cyst excision (Surgical and medical procedures) | 1/173
Sinus operation (Surgical and medical procedures) | 5/173
Aneurysm (Vascular disorders) | 2/173
Aortic stenosis (Vascular disorders) | 1/173
Arterial thrombosis (Vascular disorders) | 1/173
Arterial thrombosis limb (Vascular disorders) | 1/173
Flushing (Vascular disorders) | 3/173
Haematoma (Vascular disorders) | 5/173
Hot flush (Vascular disorders) | 5/173
Hypertension (Vascular disorders) | 27/173
Intermittent claudication (Vascular disorders) | 1/173
Pallor (Vascular disorders) | 1/173
Peripheral vascular disorder (Vascular disorders) | 1/173
Raynaud's phenomenon (Vascular disorders) | 2/173
Thrombosis (Vascular disorders) | 1/173
Vein disorder (Vascular disorders) | 1/173
Insomnia (Psychiatric disorders) | 17/173
Panic Disorder (Psychiatric disorders) | 1/173
Somnolence (Nervous system disorders) | 7/173
Neuropathy peripheral (Nervous system disorders) | 19/173
Sensory Disturbance (Nervous system disorders) | 2/173
Gingival abscess (Infections and infestations) | 1/173
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1/173
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49/173

LIMITATIONS AND CAVEATS:
Study terminated early due to business and operational issues. All subjects who were treated with inhaled insulin in parent protocols(217-102,-103,or-104) or in extension protocols (217-102E,-103E,-104E,or A2171036)are included in safety evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.